CLINICAL TRIAL: NCT06868225
Title: Prospective Study to Codify Coronary Lesions Based on Fluid Mechanics and Acoustic Mechanisms
Brief Title: Scientific Rationale and Design for a Prospective Study to Codify Coronary Lesions Based on Fluid Mechanics and Acoustic Mechanisms
Status: Not yet recruiting | Type: Observational
Sponsor: Tan Tao University, School of Medicine (Other)
Responsible Party: Principal Investigator, Thach Nguyen, Academic Dean, Tan Tao University, School of Medicine
Other Study IDs: TTU.RS.25.302.001
Record Dates: First submitted 2025-03-06; First posted 2025-03-10 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Unstable Angina (UA)
MeSH Terms: conditions — Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients coming to the cardiac catheterization laboratories for coronary angiogram: patients coming to the cardiac catheterization laboratories (CCL) for out-patient coronary angiography with diagnosis of unstable angina were screened for inclusion.

SUMMARY:
From January 2020 to June 2025, patients coming to the cardiac catheterization laboratories (CCL) for out-patient coronary angiography with diagnosis of unstable angina were screened for inclusion. Patients were included in the study if they had previously undergone one or more coronary angiograms, allowing for a longitudinal comparison of dynamic flow and phenomena between the two or more angiograms.

DETAILED DESCRIPTION:
Patients with history of prior percutaneous coronary intervention (PCI), coronary artery bypass graft surgery (CABG) were excluded. The aortic stenosis patients were also excluded if they had end-stage disease with survival time <6 months or if they had other severe hemodynamic disturbances such as hypotension from non-cardiac problems (sepsis, bleeding, etc).

ELIGIBILITY:
Inclusion Criteria: Patients were included in the study if they had one or two lesions in coronary angiograms. -

Exclusion Criteria: Patients with history of prior percutaneous coronary intervention (PCI), coronary artery bypass graft surgery (CABG) were excluded.

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all patients without prior PCI nor CABG
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
New lesion | 3 months
  If having new lesion

IPD SHARING:
Plan to Share IPD: Undecided
Will provide infos if needed